CLINICAL TRIAL: NCT03669523
Title: A Multicenter Phase II Study Evaluating Denosumab (XGEVA®) in Combination with Nivolumab (OPDIVO®) As Second-line Therapy for Patients with Stage IV Non-small-cell Lung Cancer (squamous and Non-squamous) with Bone Metastases: DENIVOS STUDY
Brief Title: Denosumab and Nivolumab Combination As 2d-line Therapy in Stage IV NSC Lung Cancer with Bone Metastases (DENIVOS)
Acronym: DENIVOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: French Lung Cancer Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P_2017_007; 2018-001105-85 (EudraCT Number)
Record Dates: First submitted 2018-09-05; First posted 2018-09-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Bone Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: National (French), multicenter, prospective, open, single-arm phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Denosumab-nivolumab combination (Experimental): Both drugs to be continued until progression or unacceptable toxicity and for a maximum of two years
  Interventions: Drug: Denosumab-nivolumab combination

INTERVENTIONS:
Drug: Denosumab-nivolumab combination — * Denosumab: 120 mg every 4 weeks subcutaneously
  * Nivolumab: 240mg intravenously on day 1 every 2 weeks

SUMMARY:
Bone metastases are common in Non-Small Cell Lung Cancer (NSCLC). They most often occur during disease progression. It is thought that more than half of the patients with bone metastases will have at least 1 skeletal-related event (SRE, i.e. pathological fractures, medullary compression, analgesic radiotherapy, preventive and/or analgesic surgery and hypercalcemia).

Expert and medical Society guidelines, notably European Society for Medical Oncology in 2014, then in 2016, recommended using anti-resorptive agents (bisphosphonates or denosumab) to prevent SREs, attenuate pain and improve the quality of life, and decrease the medical-economic impact of this major metastatic site. Denosumab was accorded marketing authorization in France in 2011 as an anti-resorptive agent for bone metastases to delay the occurrence of SREs in lung-cancer patients.

Immunotherapy, notably immune-checkpoint inhibitors, like nivolumab (anti-programed death-1), has recently become an integral part of the therapeutic arsenal against NSCLCs. Nivolumab was accorded marketing authorization based on the phase III CHECKMATE 017 (squamous cell NSCLCs) and CHECKMATE 057 (non-squamous cell NSCLCs) trials versus docetaxel, after the phase II CHECKMATE 063 trial.

The denosumab-nivolumab combination is commonly used in current practice but has not been evaluated prospectively. The aim of this trial is to evaluate the combination of denosumab and nivolumab in second line of NSCLC with bone metastases.

DETAILED DESCRIPTION:
Bone metastases are common in Non-Small Cell Lung Cancer (NSCLC), affecting 30-65% of the patients, depending on the series. They most often occur during disease progression (59.7% in the French Lung Cancer Group trial). The frequency of skeletal-related events (SREs) (pathological fractures, medullary compression, analgesic radiotherapy, preventive and/or analgesic surgery and hypercalcemia) is high. It is thought that more than half of the patients with bone metastases will have at least 1 SRE, with rates ranging from 55% to 62%.

Expert and medical Society guidelines, notably European Society for Medical Oncology in 2014, then in 2016, recommended using anti-resorptive agents (bisphosphonates or denosumab) to prevent SREs, attenuate pain and improve the quality of life, and decrease the medical-economic impact of this major metastatic site.

Denosumab is a humanized monoclonal antibody. It mimics the action of osteoprotegerin (OPG), thereby inhibiting osteoclastogenesis by blocking the binding of the receptor activator of nuclear factor-kappaB (RANK) to its ligand (RANKL), and thus interrupts the vicious circle between tumor cells and bone. RANK is a transmembrane protein expressed on osteoclasts, and its ligand, RANKL, is soluble and secreted by osteoblasts. Denosumab was accorded marketing authorization in France in 2011 as an anti-resorptive agent for bone metastases to delay the occurrence of SREs in lung-cancer patients. The results of 3 phase III studies evaluating the place of denosumab versus zoledronic acid have been published. Lung cancers were included in the trial examining solid tumors (other than breast and prostate) and multiple myeloma, and represented 40% of the population. In a non-inferiority analysis, the primary objective was reached with denosumab prolonging by approximately 4 months the time to the first SRE (20.6 versus 16.3 months, hazard ratio 0.84 [95% confidence interval 0.71-0.98] p=0.0007). In the lung-cancer subgroup, this difference did not reach significance (hazard ratio 0.85 [95% confidence interval 0.65-1.12]). In contrast, the exploratory analysis of that subgroup showed overall survival prolonged by 1.2 months for the denosumab arm versus zoledronic acid (8.9 versus 7.7 months, hazard ratio 0.8 [95% confidence interval 0.67-0.95] p=0.01).

Immunotherapy, notably immune-checkpoint inhibitors (ICPIs), like nivolumab (anti-programed death-1 (PD-1)), has recently become an integral part of the therapeutic arsenal against NSCLCs. Nivolumab was accorded marketing authorization based on the phase III CHECKMATE 017 (squamous cell NSCLCs) and CHECKMATE 057 (non-squamous cell NSCLCs) trials versus docetaxel, after the phase II CHECKMATE 063 trial. The search for a biomarker predictive of the response to immunotherapy is becoming more-and-more crucial, so as not to expose patients who risk early cancer hyper-progression. Immunohistochemical labeling of PD-1 ligand (PD-L1) on tumor cells (± infiltrating the stroma) is the most studied and reliable biomarker. Knowing its status has become indispensable in immunotherapy trials because an elevated PD-L1 has been correlated to a better response. Prescribing second-line nivolumab is not conditioned by the PD-L1 status because those trials had not foreseen stratification according to this criterion's status. However, post-hoc analysis of PD-L1 in the CHECKMATE 057 trial on non-squamous cell NSCLCs showed prolonged overall survival for patients with PD-L1-positive tumors, whether the positivity threshold was 1%, 5% or 10%. Thus, knowing the PD-L1 status is necessary to interpret the results of immunotherapy trials.

The RANK-RANKL system was studied in preclinical osteoimmunology models. It is expressed by certain cells, notably antigen-presenting cells, such as dendritic cells or lymphocytes, essential for the adaptive immunity function solicited by immunotherapy. It is part of the tumor necrosis factor receptor (TNF-R) family and is implicated in the interactions between dendritic cells and lymphocytes. The RANK-RANKL role in the development and function of regulatory T cells (Tregs) remains poorly elucidated. Information on the interaction of the RANK-RANKL system and adaptive immunity obtained with the preclinical models is discordant and rare. A case report on a patient with melanoma bone metastases treated with denosumab and ipilimumab (ICPI of the anti-cytotoxic T-lymphocyte antigen 4 type) obtained a promising carcinological outcome, without any sign of deleterious interaction.

The aim of this trial is to evaluate the combination of denosumab and nivolumab in second line of NSCLC with bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically proven stage IV NSCLC
* Patients who had received first-line platin salt-based chemotherapy and will be given second-line nivolumab;
* Patients with bone metastases, symptomatic or not, confirmed by X-rays, CT scan, MRI, PET-CT scan or technetium bone scintigraphy
* Presence of at least 1 measurable target lesion, according to RECIST criteria 1.1, in a non-irradiated site
* For non-squamous cell NSCLC, patients without known activating epidermal growth factor receptor mutation, anaplastic lymphoma kinase (ALK) or reactive oxygen species (ROS)-1 translocation, or B-Raf proto-oncogene, serine/threonine kinase (BRAF V600) mutation
* PD-L1 status known and expressed as a percentage of tumor cells; assessed at the diagnosis or the more recent PD-L1 expression status available.
* Eastern Cooperative Oncology Group Performance Status 0/1
* Estimated life-expectancy ≥12 weeks
* No prior malignant tumor during the previous 5 years, except for in situ carcinomas of the cervix or basal or squamous cell carcinomas of the skin adequately treated;
* Adequate organ function determined by laboratory analyses less than 7 days before inclusion:

  * Normal hepatic function: bilirubin < 1.5× normal (N), alanine aminotransferase and aspartate aminotransferase <2.5× N or <5× N if hepatic metastases are present
  * Renal function (renal clearance of creatinine at least ≥45 mL/min)
  * Hematological function: absolute number of neutrophils ≥1.5×109/L and/or platelets ≥100×109/L, hemoglobin ≥8 g/dL
* Women of child-bearing age must use an effective contraceptive method and mechanical contraception during and up to 6 months after the end of treatment;
* Men must use effective contraception during and up to 6 months after the treatment period
* Patient with asymptomatic brain metastases (treated or not) OR symptomatic brain metastases but adequately treated and controlled at the time of enrolment (without or with corticotherapy ≤ 10mg/day), can be included. Carcinomatous meningitis is excluded regardless of clinical stability
* Subjects must have signed and dated an approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
* Patient affiliated or benefitting from the French national health insurance program

Exclusion Criteria:

* Patients previously treated with immunotherapy
* Patients with symptomatic cerebral metastases not treated and not controlled
* Contraindication to nivolumab use:

  * Prior autoimmune disease(s), define as disease required systemic treatment in the past (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
  * Prior diffuse interstitial pneumopathy
  * Systemic immunosuppressive therapy; define as steroid medication at a dose greater than prednisone 10 mg/day or equivalent. For patients with mismatch repair-deficient high-grade gliomas, concurrent steroid medication at a dose greater than prednisone 20mg/day or equivalent
* Contraindication for denosumab use:

  * Poor dental status requiring immediate specialized management, like oral surgery
  * Prior or current signs of osteonecrosis of the jaw/osteomyelitis
  * Invasive dental intervention schedule during the study or not yet healed
* Patient with known sensitivity to any of the products to be administered during the study
* Concomitant administration of bisphosphonates
* Hypocalcemia or severe uncorrected hypercalcemia
* Medical or psychological condition preventing informed consent
* Pregnant or breastfeeding woman
* PD-L1-status results unavailable
* Simultaneous participation of the patient in another clinical research trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) according to the PD-L1-expression rate (threshold set at 1%) | At 24 months
  ORR (Complete and Partial Responses) will be expressed as number, percentage and 95% confidence interval, calculated with the exact method.
  The evaluation of ORR, according to PD-L1-expression rate, using RECIST criteria 1.1, will be performed by the investigator in each center. A panel of French Lung Cancer Group investigators meeting 3 times/year will then validate it by a second reading.

SECONDARY OUTCOMES:
Disease-control rate (DCR) | up to 24 months
  The DCR (complete and partial responses + stabilized disease using RECIST criteria 1.1) will be expressed as number, percentage and 95% confidence interval, calculated with the exact method, for the entire population, then by subgroups according to the PD-L1-expression rate, and histological type (adenocarcinoma versus squamous-cell).
Overall survival | over 24 months
  Overall survival over 24 months will be described using the Kaplan-Meier method. Log-rank tests will be used to analyze subgroups according to PD-L1-expression rate, then histological type (adenocarcinoma versus squamous-cell). Survival medians, in the overall population and according to PD-L1-expression rate, then histological type (adenocarcinoma versus squamous-cell) will be calculated.
Progression-free survival | over 24 months
  Progression-free survival over 24 months will be described with the Kaplan-Meier method. Log-rank tests will be used to analyze subgroups according to PD-L1-expression rate, then histological type (adenocarcinoma versus squamous-cell). Progression-free survival medians, in the overall population and according to PD-L1-expression rate, then histological type (adenocarcinoma versus squamous-cell) will be calculated.
Overall Response Rate for the entire population | At 24 months
  The 24-month Overall Response Rate (Complete and Partial Responses using RECIST criteria 1.1) for the entire population, then according to histological type (adenocarcinoma versus squamous-cell) will be expressed as number, percentage and 95% confidence interval, calculated with the exact method.
Overall Response Rate according to the histological type (adenocarcinoma versus squamous cell) | At 24 months
  The 24-month Overall Response Rate (Complete and Partial Responses using RECIST criteria 1.1) for the entire population, then according to histological type (adenocarcinoma versus squamous-cell) will be expressed as number, percentage and 95% confidence interval, calculated with the exact method.
Time to the first Skeletal-Related Event in months | Over 24 months
  The time to an Skeletal-Related Event will be estimated with the Kaplan-Meier method over 24 months of follow-up.
  Skeletal-Related Event are defined as pathological fractures, medullary compression, analgesic radiotherapy, preventive and/or analgesic surgery and hypercalcemia.
Incidence of adverse events, serious adverse events, deaths and biological abnormalities | up to 24 months
  Scored according to NCI CTCAE V4.0 terminology

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Decroisette, MD, Principal Investigator — CH Annecy Genevois
Locations (27):
- France (27):
  - CH du Pays d'Aix, Aix-en-Provence
  - Chu Angers, Angers
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - CHU Morvan - Institut de Cancérologie et d'Hématologie, Brest
  - CH Intercommunal, Créteil
  - Ch Intercommunal Elbeuf Louvier Val de Reuil, Elbeuf
  - CH Intercommunal des Alpes du Sud, Gap
  - Hôpital Robert Boulin, Libourne
  - Chu Dupuytren, Limoges
  - CH Marne La Vallée, Marne La Vallée
  - Hopital Européen, Marseille
  - Hopital Nord APHM, Marseille
  - CH Meaux, Meaux
  - Centre Catalan d'Oncologie, Perpignan
  - CH Annecy-Genevois, Pringy
  - CHU Hôpital Pontchailloux, Rennes
  - CHU Rouen, Rouen
  - CHU La Réunion - Site de Bellepierre, Saint-Denis
  - Groupe Hospitalier Sud Réunion - CHU de la Réunion, Saint-Pierre
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CLCC Paul Strauss, Strasbourg
  - Centre Hospitalier de Bigorre, Tarbes
  - Hôpital d'Instruction des Armées Saint-Anne, Toulon
  - CHITS Toulon Sainte-Musse, Toulon
  - Hôpital André Mignot Centre Hospitalier de Versailles, Versailles
  - CH Villefranche sur Saone, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Undecided